CLINICAL TRIAL: NCT00920023
Title: Improved Pre-Operative Staging of Pancreatic Cancer Using Superparamagnetic Iron Oxide Magnetic Resonance Imaging (SPIO MRI)
Brief Title: Pre-Operative Staging of Pancreatic Cancer Using Superparamagnetic Iron Oxide Magnetic Resonance Imaging (SPIO MRI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ralph Weissleder, MD, Professor of Radiology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-085
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Pancreatic Cancer
Keywords: SPIO MRI; Feridex
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ferumoxtran-10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SPIO MRI (Experimental)
  Interventions: Drug: Superparamagnetic Iron Oxide Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Superparamagnetic Iron Oxide Magnetic Resonance Imaging — Two MRIs will be performed over a two day period. The second scan will be done 48 hours after intravenous infusion of ferumoxytol
  Other Names: SPIO MRI; USPIO; Feruoxytol

SUMMARY:
The purpose of this research study is to see if a specific kind of MRI, called Ultrasmall Superparamagnetic Iron Oxide Magnetic Resonance Imaging (USPIO MRI), which uses an FDA-approved therapeutic agent(Feraheme) to see if it is able to identify small and otherwise undetectable lymph node metastases in people who have pancreatic cancer and are scheduled for surgical resection.

DETAILED DESCRIPTION:
* On the first day, study participants will undergo 2 MRI examinations. A scan will be done prior to administration of the contrast agent (Feraheme) and then a second scan immediately after administration. On the second day, study participants will be asked to return for a third MRI.
* All MRI scans will be done at Massachusetts General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Locally resectable pancreatic mass present on one or more pre-operative imaging modalities
* Must demonstrate no evidence of distant metastases as assessed by chest/abdomen/pelvis CT scan
* Deemed eligible for resection with curative intent by a treating surgeon who is listed as an investigator on this study
* 18 years of age or older
* No uncontrolled serious medical or psychiatric illness
* Women of childbearing potential must not be pregnant or lactating

Exclusion Criteria:

* Known allergy to iron or dextran
* Pregnant or lactating
* Counter-indication to MRI, such as the presence of metallic prostheses or implanted metal device
* Sickle cell disease or hemoglobinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-07; Primary Completion 2012-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Weissleder, MD, PhD, Principal Investigator — Massachussetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SPIO MRI: Superparamagnetic Iron Oxide Magnetic Resonance Imaging: Three MRIs will be performed over a two day period. The second scan will be done 48 hours after intravenous infusion of ferumoxytol
Period: Overall Study
Arm/Group | SPIO MRI
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SPIO MRI
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Sensitivity High Resolution Magnetic Resonance Imaging With Lymphotrophic Superparamagnetic Nanoparticles to Identify Small and Otherwise Undetectable Lymph Node Metastases.
Description: Using Pathology as the gold standard the excised nodes were correlated and the percentage of positive cases were measured on the post contrast exam. Sensitivity is the percentage of positive cases (i.e., metastases confirmed using pathology) identified as positive.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of positive cases
Arm/Group | SPIO MRI
Number analyzed (Participants) | 15
percentage of positive cases | 83.3 [36.4 to 99.1]

2. Primary Outcome: To Determine the Specificity of High Resolution Magnetic Resonance Imaging With Lymphotrophic Superparamagnetic Nanoparticles to Identify Small and Otherwise Undetectable Lymph Node Metastases.
Description: Using Pathology as the gold standard the excised nodes were correlated and the percentage of true negative nodes were measured on the post contrast exam. Specificity is the percentage of true negative cases as identified as negative.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: Percentage of true negative sample
Arm/Group | SPIO MRI
Number analyzed (Participants) | 15
Percentage of true negative sample | 80 [29.8 to 98.9]

ADVERSE EVENTS:
Arm/Group | SPIO MRI
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No